CLINICAL TRIAL: NCT00696189
Title: The Effects of Nitrous Oxide on Intraocular Pressure and Ocular Perfusion
Brief Title: Effects of Nitrous Oxide on Intraocular Pressure
Status: Terminated | Type: Observational
Why Stopped: PI is no longer at this institution
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 0120060249; 0120060249
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Post Operative Visual Loss
Keywords: Post operative visual loss (POVL); Intraocular pressure (IOP); Nitrous oxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The concept of ocular perfusion pressure (OPP), is defined as the difference between the mean arterial pressure (MAP) and the intraocular pressure (IOP.)It has been hypothesized that unopposed decreases in MAP, increases in IOP or a combination of the two may result in hypo perfusion of the eye and can cause an ocular infarction at the level of the retina or optic nerve, leading to varying degrees of visual loss which is frequently bilateral and irreversible.

Both the prone position and downward head tilting (Trendelenburg position) have been associated with increases in IOP compared to the supine horizontal position (2,4,5,6), but it is not known whether the Trendelenburg position during surgery and anesthesia is associated with POVL.

DETAILED DESCRIPTION:
Our preliminary Phase I studies using awake volunteers confirmed the increase in IOP associated with the prone position which is attenuated, although not eliminated, with a 15 cm head up table elevation. In addition we found evidence of retinal vascular changes consistent with venous congestion over a one hour period in the prone position in five awake volunteers using digital retinal imaging.

It is known that general anesthesia decreases IOP. A critical element, however, which has not been definitively studied is the effect of individual anesthetics, specifically nitrous oxide, on IOP. It is known that nitrous oxide does increase IOP when inert gases are injected into the vitreous for treatment of retinal detachment and this phenomenon can last up to six weeks, resulting in permanent vision loss with its use. It has also been shown that nitrous oxide increases intracranial pressure (ICP,9) although this effect may be attenuated by narcotics and additional intravenous anesthetic agents. It also increases cerebral metabolic rate, potentially aggravating any compromise in blood flow. Several studies showed a significant association between elevated IOP and ICP. Therefore, it is critical to attempt to isolate the effect of nitrous oxide on IOP. Because nitrous oxide is used as an adjunct to other anesthetics, it is the most frequently used of all the inhalation anesthetics and delineating its effect on this variable will help clinicians decide whether the advantage of its use outweighs the risk.

Because general anesthesia decreases IOP and there is significant variation between subjects this study is planned using a within subject design. Patients undergoing open gynecological procedures such as hysterectomies and patients undergoing orthopedic surgery are ideal candidates for the proposed study for the following reasons. The majority of patients undergoing general anesthesia in University Hospital operating rooms require frequent table position changes which might affect the results. Therefore, we choose to study patients who will remain in one position for the majority of the operation. The hysterectomy patients offer a unique benefit because It would also be advantageous to study patients in a position known to increase IOP in order to better detect differences in anesthetic regimen and isolate the effects of a specific agent. In addition, patients undergoing orthopedic surgery such as hand and ankle procedures are commonly in a fixed supine position for the predominance of the operation. University Hospital conducts a considerably greater number of orthopedic cases than gynecological cases daily which allows for greater ease in patient enrollment. Measuring IOP in the supine Trendelenburg position offers significant technical and logistical advantages compared to the prone position and therefore taking our measurements in this position is desirable.

ELIGIBILITY:
Inclusion Criteria:

* If I am between the ages of 18 and 65 years of age and mentally capable of giving consent.
* If I am scheduled for gynecological surgery and will be placed in the Trendelenburg position (head lower than my waist) on the operating room table.

Exclusion Criteria:

* If I fail/refuse to provide an informed consent
* If I have a history of stroke or trans-ischemic attack (TIA).
* If I have a history of corneal disease.
* If I a have a sensitivity to eye drops called proparacaine
* If I have had a previous diagnosis of carotid disease.
* If I have a history of glaucoma
* If I am taking medications which may affect the pressure in my eyes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ages of 18 and 65 years of age and mentally capable of giving consent. Scheduled for gynecological surgery and will be placed in the Trendelenburg position (head lower than my waist) on the operating room table.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geordie Grant, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ, Newark, New Jersey, United States